CLINICAL TRIAL: NCT02597283
Title: A Prospective, Multi-center, Randomized Trial Comparing Biguard Stent With Regular Sirolimus-eluting Stent System for Patients With Coronary Bifurcation Lesions
Brief Title: Coronary Bifurcation Lesions Treated With Biguard Stent System
Acronym: BIGUARD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Director of Cardiology and Cath Lab, Vice President of Nanjing First Hospital, Nanjing Medical University, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFHMU20150902
Record Dates: First submitted 2015-11-02; First posted 2015-11-05 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease
Keywords: Bifurcation lesions; Percutaneous coronary intervention; Randomized controlled trial
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biguard stent system (Experimental): PCI with Biguard sirolimus-eluting bifurcation stent system
  Interventions: Device: Biguard sirolimus-eluting bifurcation stent system
- Sirolimus-eluting stent system (Active Comparator): PCI with regular sirolimus-eluting stent system
  Interventions: Device: Sirolimus-eluting stent system

INTERVENTIONS:
Device: Biguard sirolimus-eluting bifurcation stent system — PCI with Biguard sirolimus-eluting bifurcation stent system
  Other Names: Biguard Stent System
  Arms: Biguard stent system
Device: Sirolimus-eluting stent system — PCI with sirolimus-eluting stent system
  Other Names: SES
  Arms: Sirolimus-eluting stent system

SUMMARY:
This study is designed to test the hypothesis that the Biguard stent system will lead to fewer target lesion failure compared to regular stent system in patients with coronary bifurcation lesions at one year.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to compare the effect of Biguard bifurcation stent system and regular stent system in patients with bifurcation lesions. Based on the previous studies, the rate of 1-year target lesion failure was around 12% after PCI with regular stent system. And the investigators previous data showed that this event at 12-month after Biguard bifurcation stent system was 4%. Considering the lost to follow-up, it is anticipated that up to 400 patients will be enrolled in the trial. All patients will have repeat angiography at 13 months, with clinical follow-up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be age≥18 years;
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed;
* Subject is eligible for percutaneous coronary intervention (PCI);
* Subject has symptomatic coronary artery disease or documented silent ischemia;
* Subject is willing to comply with all protocol-required follow-up evaluations;
* Target lesion must be a de novo true bifurcation lesions located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.50 mm and ≤4.00 mm;
* Target lesion must have visually estimated stenosis ≥50%;
* The lesion length of main branch vessel must measure <40 mm, and the lesion length of side branch vessel must measure <20 mm (by visual estimate);
* Subject with no more than one lesion existing in the same vessel can be chosen, when several bifurcation lesions existing simultaneously;
* Subject with knowledge of trial purpose, informed consents and volition of undergoing coronary angiography and clinical follow-up voluntarily.

Exclusion Criteria:

* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute MI within two weeks;
* Subject is on dialysis or has serum creatinine level >3.0 mg/dL;
* Subject has known allergy to the study stent system or protocol-required concomitant medications;
* Subject has any other serious medical illness that may reduce life expectancy to less than 12 months; Patient with cardiac heart failure (above New York Heart Association (classification) III), or left ventricular ejection fraction (LVEF)< 30%;
* Subject with hemorrhagic tendency or history of active peptic ulcers, cerebral hemorrhage, or subarachnoid hemorrhage, cerebral stroke within half a year, as well as patients who have contraindication to anti-platelet agents or anticoagulant treatment;
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint or intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure;
* Subject Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk- Subject has more than 1 lesion that requires treatment during the index procedure;
* Target lesion meets any of the following criteria:

  1. Thrombus, or possible thrombus, present in the target vessel;
  2. Excessive tortuosity proximal to or within the lesion;
  3. Excessive angulation proximal to or within the lesion;
  4. Chronic total occlusion lesion in target vessel not re-canalized;
  5. severe calcification with unsuccessfully pre-dilated;
  6. restenosis disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Ischemia Driven Target Lesion Failure (ID-TLF) | 12 months
  The number of participants with adverse events that are related to treatment. Adverse events included cardiac death (death in which a cardiac cause cannot be excluded), Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI and Ischemia-driven target vessel revascularization (TVR) by CABG or PCI.

SECONDARY OUTCOMES:
In-stent late lumen loss in millimeter | 13 months
  In-stent MLD post-procedure minus in-stent MLD at follow-up (in-stent defined as within the margins of the stent)
Proximal Late Loss in millimeter | 13 months
  Proximal Minimum Lumen Diameter (MLD) post-procedure minus proximal MLD at follow-up (proximal defined as within 5 mm of healthy tissue proximal to stent placement)
Distal Late Loss in millimeter | 13 months
  Distal MLD post-procedure minus distal MLD at follow-up (distal defined as within 5 mm of healthy tissue distal to stent placement)
Incidence of Target Vessel Failure (TVF) | 30 days
  The number of participants with adverse events that are related to treatment. Adverse events included cardiac death (death in which a cardiac cause cannot be excluded), Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI and Ischemia-driven target vessel revascularization (TVR) by CABG or PCI.
Incidence of Target Vessel Failure (TVF) | 1 year
  The number of participants with adverse events that are related to treatment. Adverse events included cardiac death (death in which a cardiac cause cannot be excluded), Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI and Ischemia-driven target vessel revascularization (TVR) by CABG or PCI.
Incidence of Target Vessel Failure (TVF) | 3 year
  The number of participants with adverse events that are related to treatment. Adverse events included cardiac death (death in which a cardiac cause cannot be excluded), Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI and Ischemia-driven target vessel revascularization (TVR) by CABG or PCI.
Incidence of Target Vessel Failure (TVF) | 5 year
  The number of participants with adverse events that are related to treatment. Adverse events included cardiac death (death in which a cardiac cause cannot be excluded), Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI and Ischemia-driven target vessel revascularization (TVR) by CABG or PCI.
Incidence of Ischemia Driven Target Lesion Revascularization (ID-TLR) | 30 days
  The number of participants with revascularization at target lesion associated with any of following: functional ischemia study Ischemic symptoms & angiographic diameter stenosis ≥50% by core lab quantitative coronary angiography (QCA), revascularization of a target lesion with angiographic diameter stenosis ≥70% by core laboratory QCA without angina or functional study.
Incidence of Ischemia Driven Target Lesion Revascularization (ID-TLR) | 1 year
  The number of participants with revascularization at target lesion associated with any of following: functional ischemia study Ischemic symptoms & angiographic diameter stenosis ≥50% by core lab quantitative coronary angiography (QCA), revascularization of a target lesion with angiographic diameter stenosis ≥70% by core laboratory QCA without angina or functional study.
Incidence of Ischemia Driven Target Lesion Revascularization (ID-TLR) | 3 year
  The number of participants with revascularization at target lesion associated with any of following: functional ischemia study Ischemic symptoms & angiographic diameter stenosis ≥50% by core lab quantitative coronary angiography (QCA), revascularization of a target lesion with angiographic diameter stenosis ≥70% by core laboratory QCA without angina or functional study.
Incidence of Ischemia Driven Target Lesion Revascularization (ID-TLR) | 5 year
  The number of participants with revascularization at target lesion associated with any of following: functional ischemia study Ischemic symptoms & angiographic diameter stenosis ≥50% by core lab quantitative coronary angiography (QCA), revascularization of a target lesion with angiographic diameter stenosis ≥70% by core laboratory QCA without angina or functional study.
Incidence of Ischemia Driven Target Vessel Revascularization (ID-TVR) | 30 days
  The number of participants with revascularization at the target vessel associated with any of the following Positive functional ischemia study Ischemic symptoms and angiographic diameter stenosis ≥ 50% by core laboratory QCA Revascularization of a target vessel with angiographic diameter stenosis ≥ 70% by core laboratory QCA without angina or positive functional study Derived from Non-Hierarchical Subject Counts of Adverse Events
Incidence of Ischemia Driven Target Vessel Revascularization (ID-TVR) | 1 year
  The number of participants with revascularization at the target vessel associated with any of the following Positive functional ischemia study Ischemic symptoms and angiographic diameter stenosis ≥ 50% by core laboratory QCA Revascularization of a target vessel with angiographic diameter stenosis ≥ 70% by core laboratory QCA without angina or positive functional study Derived from Non-Hierarchical Subject Counts of Adverse Events
Incidence of Ischemia Driven Target Vessel Revascularization (ID-TVR) | 3 year
  The number of participants with revascularization at the target vessel associated with any of the following Positive functional ischemia study Ischemic symptoms and angiographic diameter stenosis ≥ 50% by core laboratory QCA Revascularization of a target vessel with angiographic diameter stenosis ≥ 70% by core laboratory QCA without angina or positive functional study Derived from Non-Hierarchical Subject Counts of Adverse Events
Incidence of Ischemia Driven Target Vessel Revascularization (ID-TVR) | 5 year
  The number of participants with revascularization at the target vessel associated with any of the following Positive functional ischemia study Ischemic symptoms and angiographic diameter stenosis ≥ 50% by core laboratory QCA Revascularization of a target vessel with angiographic diameter stenosis ≥ 70% by core laboratory QCA without angina or positive functional study Derived from Non-Hierarchical Subject Counts of Adverse Events
Incidence of Ischemia Driven Major Adverse Cardiac Event (MACE) | 30 days
  The number of participants with adverse events that are related to treatment. Adverse events comprised of cardiac death, Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI.
Incidence of Ischemia Driven Major Adverse Cardiac Event (MACE) | 1 year
  The number of participants with adverse events that are related to treatment. Adverse events comprised of cardiac death, Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI.
Incidence of Ischemia Driven Major Adverse Cardiac Event (MACE) | 3 year
  The number of participants with adverse events that are related to treatment. Adverse events comprised of cardiac death, Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI.
Incidence of Ischemia Driven Major Adverse Cardiac Event (MACE) | 5 year
  The number of participants with adverse events that are related to treatment. Adverse events comprised of cardiac death, Myocardial infarction (MI, classified as Q-wave and non-Q wave), Ischemia-driven target lesion revascularization (TLR) by CABG or PCI.
In-stent % Angiographic Binary Restenosis (% ABR) Rate | 13 months
  Percent of subjects with a follow-up in-stent percent diameter stenosis of ≥ 50% per quantitative coronary angiography (QCA)
In-segment % Angiographic Binary Restenosis (% ABR) Rate | 13 months
  Percent of subjects with a follow-up in-segment percent diameter stenosis of ≥ 50% per quantitative coronary angiography (QCA)

OTHER OUTCOMES:
Acute Success: Clinical Procedure | 7 days
  Successful delivery and deployment of study stent/s @ the intended target lesion and successful withdrawal of the stent delivery system with final residual stenosis < 50%.
Acute Success: Clinical Device | 7 days
  Successful delivery and deployment of 1st implanted study stent/s @ the intended target lesion and successful withdrawal of the stent delivery system with final residual stenosis < 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Principal Investigator — Director of Cardiology and Cath Lab, Nanjing First Hospital

IPD SHARING:
Plan to Share IPD: No